CLINICAL TRIAL: NCT07064889
Title: The Combination of Oral Upadacitinib and High-dose Dexamethasone vs High-dose Dexamethasone as First-line Treatment in Adult Immune Thrombocytopenia: A Multicenter, Randomized, Open-label Trial
Brief Title: The Combination of Upadacitinib and High-dose Dexamethasone as First-line Treatment in Adult Immune Thrombocytopenia
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Collaborators: Beijing Hospital (Other Government); Navy General Hospital, Beijing (Other); Beijing Aerospace General Hospital (Other); Qilu Hospital of Shandong University (Other); Beijing Tongren Hospital (Other)
Responsible Party: Principal Investigator, Xiao Hui Zhang, Vice president of Peking Univeristy Institute of Hematology, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ITP-UPA-001
Record Dates: First submitted 2025-07-07; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Dexamethasone; upadacitinib

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Upadacitinib and HD-DXM (Experimental): Dexamethasone 40 mg per day, 4 consecutive days (the 4-day course of dexamethasone was repeated in the case of lack of response by day 10) and Upadacitinib 15mg qd po, 12 consecutive weeks
  Interventions: Drug: Dexamethasone; Drug: Upadacitinib
- HD-DXM (Active Comparator): Dexamethasone 40 mg per day, 4 consecutive days (the 4-day course of dexamethasone was repeated in the case of lack of response by day 10)
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone, 40 mg/d, for 4 days (The 4-day course of dexamethasone was repeated in the case of lack of response by day 10)
Drug: Upadacitinib — Upadacitinib 15mg qd for 12 weeks
  Arms: Upadacitinib and HD-DXM

SUMMARY:
Randomized, open-label, multicenter study to compare the efficacy and safety of Upadacitinib plus high-dose dexamethasone compared to high-dose dexamethasone monotherapy for the first-line treatment of adults with primary immune thrombocytopenia (ITP).

DETAILED DESCRIPTION:
The investigators are undertaking a parallel group, multicenter, randomized controlled trial of adults ITP patients in China. Patients were randomized to Upadacitinib + high-dose dexamethasone and high-dose dexamethasone monotherapy group. Platelet count, bleeding and other symptoms were evaluated before and after treatment. Adverse events are also recorded throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed newly-diagnosed, treatment-naive ITP;
2. Platelet counts <30×109/L ;
3. Platelet counts < 50×109/L and significant bleeding symptoms (WHO bleeding scale 2 or above);
4. Willing and able to sign written informed consent.

Exclusion Criteria:

1. Received chemotherapy or anticoagulants or other drugs affecting the platelet counts within 6 months before the screening visit;
2. Received first-line and second-line ITP-specific treatments (eg, steriods, cyclophosphamide, 6-mercaptopurine, vincristine, vinblastine, etc) ;
3. Current HIV infection or hepatitis B virus or hepatitis C virus infections;
4. Active infection;
5. Maligancy;
6. Severe medical condition (lung, hepatic or renal disorder) other than chronic ITP. Unstable or uncontrolled disease or condition related to or impacting cardiac function (e.g., unstable angina, congestive heart failure, uncontrolled hypertension or cardiac arrhythmia);
7. Female patients who are nursing or pregnant, who may be pregnant, or who contemplate pregnancy during the study period; a history of clinically significant adverse reactions to previous corticosteroid therapy
8. Have a known diagnosis of other autoimmune diseases, established in the medical history and laboratory findings with positive results for the determination of antinuclear antibodies, anti-cardiolipin antibodies, lupus anticoagulant or direct Coombs test;
9. Patients who are deemed unsuitable for the study by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2025-07-30 (Estimated); Primary Completion 2027-07-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Sustained response | 6 month
  The maintenance of platelet count ≥ 30 x 10^9/L, at least 2-fold increase of the baseline count, the absence of bleeding, and no need for rescue medication at the 6-month follow-up.

SECONDARY OUTCOMES:
complete response (CR) | day 14
  complete response (CR) was defined as platelet count more than 100,000 per cubic millimeter and absence of bleeding
Response (R) | day 14
  Response (R) as platelet count more than 30,000 per cubic millimeter and at least 2-fold increase of the baseline count and absence of bleeding.
Number of patients with bleeding | 6 month
  Number of patients with bleeding complication ( WHO bleeding score).
Number of patients with adverse events | 6 month
  Number of patients with adverse events
Time to response | 6 month
  The time from starting treatment to time of achievement of CR or R
Duration of response (DOR) | 6 month
  Duration of response at 6-month follow up
Loss of response | 6 month
  Platelet counts below 100 x 109/L or bleeding (from CR) or platelet counts below 30 x 109/L, less than 2-fold increase of baseline platelet count or bleeding (from R)
Health related quality of life | 6 month
  Health-related quality of life using the Immune Thrombocytopenic Purpura-Patient Assessment Questionnaire (ITP-PAQ)

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to data, including deidentified individual participant data, and the study protocol from this clinical trial. These data will be available beginning 3 months and ending 36 months following publication. All requests must include a description of the research proposal and be sent to the corresponding author (zhangxh@bjmu.edu.cn). Data requestors will need to sign a data access agreement to obtain access.
Supporting Information: Study Protocol, SAP
Time Frame: These data will be available beginning 3 months and ending 36 months following publication.
Access Criteria: All requests must include a description of the research proposal and be sent to the corresponding author (zhangxh@bjmu.edu.cn). Data requestors will need to sign a data access agreement to obtain access.